CLINICAL TRIAL: NCT05357313
Title: A Randomized Placebo-controlled Trial for Adjunctive Bright Light Therapy in Patients With Bipolar Depression and Eveningness
Brief Title: Adjunctive Bright Light Therapy in Patients With Bipolar Depression and Eveningness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Joey WY Chan, Clinical Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020.676T; 14111502 (Other Grant/Funding Number: General Research Fund (GRF), Research Grants Council, University Grant Committee)
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Bipolar Depression
Keywords: Bipolar depression; Eveningness; Bright light therapy
MeSH Terms: conditions — Bipolar Disorder | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The subjects will be explained that the study aims to test the efficacy of the different modalities of non-pharmacological treatments for depression including bright light therapy and the negative ion generator, without mentioning which one is the placebo. An independent outcome assessor will be blinded to the treatment allocation throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright light therapy group (Experimental): 10,000lux bright light
  Interventions: Device: Bright light therapy
- Placebo group (Placebo Comparator): inactive negative ion generator
  Interventions: Device: Inactive negative ion generator

INTERVENTIONS:
Device: Bright light therapy — Exposure to 10,000lux bright light for 30minutes a day for six weeks
  Arms: Bright light therapy group
Device: Inactive negative ion generator — Exposure to an inactive negative ion generator for 30 minutes a day for six weeks
  Arms: Placebo group

SUMMARY:
This is a randomized placebo-controlled trial to examine the efficacy of six-week bright light therapy as adjunctive treatment for patient with bipolar depression and eveningness.

DETAILED DESCRIPTION:
This randomized placebo-controlled trial aims to evaluate the efficacy of adjunctive BLT in addition to their maintenance treatment in reducing depressive symptoms. The second aim of the study is to explore the effects of BLT on sleep-wake changes and the sleep disturbances.

Method: Each eligible participant will be randomized to either i) bright light therapy (BLT) or ii) inactive negative ion generator (placebo) treatment for 30-minutes daily at their habitual wake time for a total of six weeks. Participants will be evaluated at baseline, 2nd, 4th and 6th week for depression and insomnia symptoms. Actigraphy will be done at baseline and in the last week of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years.
2. Is capable to give informed consent.
3. Meeting the diagnostic criteria of bipolar depression (including both bipolar I and II disorders) by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V), Disorders (SCID-V).
4. a score 20 or above representing current moderate or severe episode of major depression and a score of at least 1 on items H1 or H2 on the Structured Interview Guide for the Hamilton Depression Rating Scale with Atypical Depression Supplement (SIGH-ADS), corresponding to at least moderate severity.
5. A score of 41 or less by the Morningness-Eveningness Questionnaire which represents eveningness.
6. On a stable dose of antimanic treatment for bipolar disorder for at least four weeks.

Exclusion Criteria:

1. Major Depressive Disorder fulfilling the Seasonal Pattern Specifier of the DSM-V (Seasonal Affective Disorder).
2. A past history of rapid-cycling within the past twelve months or a Young Mania Rating Scale more than 12 at screening
3. A current or past history of schizophrenia, mental retardation, organic mental disorder; or current substance use disorder.
4. Presence of psychotic symptoms or substantial suicidal risk as judged by the clinician and/or screening instruments.
5. Presence of contraindications to bright light therapy: for example, history of light induced migraine/ epilepsy; current use of photosensitizing medications such as St. John's wart; presence of eye disease: e.g. retinal blindness, severe cataract, glaucoma, and photosensitive skin condition e.g. systemic lupus erythematosus
6. Significant medical condition/ hearing impairment/ speech deficit leading to incapability of completing clinical interview.
7. Regular shift-workers or trans-meridian flight in the past 3 months or during study
8. Enrolment in another clinical trial of an investigational medicinal product or device.
9. Receiving regular psychotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change of depressive symptoms score | at the end of treatment
  Change in the score of the Structural Interview Guide for the Hamilton Depression Rating Scale with atypical depression supplement (SIGH-ADS), SIGH-ADS scores range from 0-79; higher score indicates greater depression severity.

SECONDARY OUTCOMES:
Change of insomnia symptoms | at the end of treatment
  The change in the score of the Insomnia Severity Index (ISI), which ranges from 0-28, higher score indicates higher severity of insomnia

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No